CLINICAL TRIAL: NCT06204172
Title: Intensive Neurowave Emotional Stimulation (INES): A Pioneering RCT Investigating Cognitive-Motor Impact in Consciousness Disorders Post Severe Brain Injury
Brief Title: Intensive Neurowave Emotional Stimulation (INES)
Acronym: INES_ABI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Maria Grazia Maggio, Principal Investigator, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02/2023
Record Dates: First submitted 2023-12-15; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Disorders of Consciousness
Keywords: Multisensory Stimulation; Acquired Brain Injury; Cognitive-Motor rehabilitation; Disorders of Consciousness; Metabolic-Nutritional Status
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries

STUDY DESIGN:
Intervention Model Description: The study adopts a Randomized Controlled Pilot design, an interventional, non-pharmacological, monocentric approach, aiming to explore cognitive-motor effects using advanced multisensory stimulation, the Neurowave system. Enrollment of at least 20 eligible subjects will occur consecutively at the Neurorehabilitation Unit of Piedmont Hospital. The study entails comprehensive baseline assessments (T0), succeeded by a one-month intensive cycle of advanced multisensory training. The experimental group will undergo Neurowave (INES) stimulation, while the control group will receive conventional multisensory stimulation (ISES - Intensive Sensorial Emotional Stimulation) without the advanced technological tool. Evaluations after each training cycle (T1) and a one-month follow-up (T2) will yield insights into short-term and long-term outcomes encompassing clinical-psychometric, neurophysiological, and metabolic-nutritional dimensions.
Who Masked: Participant, Investigator
Masking Description: To minimize the effect of selection bias (or even selection distortion), subject enrollment in the respective study arms (experimental or control) will be carried out through simple randomization sampling, i.e., randomly. Randomization is achieved by extracting numbers from a list, referred to as the 'sampling list,' which includes all individuals in the study population
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): patients will receive Neurowave multisensory stimulation with concurrent event-related potential acquisition. This intensive training spans five days a week over four weeks, with each session lasting 45 minutes, summing up to 20 sessions. During each session, participants will encounter personalized visual and auditory stimuli. Neurowave treatment comprises an intensive intervention, presenting emotionally significant audio-visual content linked to the patient's life history. Within Neurowave use, visual stimuli will be complemented by primary auditory stimulation, involving exposure to emotionally charged everyday sounds.
  Interventions: Device: Intensive Neurowave Emotional Stimulation (INES)
- Control group (Active Comparator): Participants will receive primary auditory stimulation featuring familiar and emotionally evocative everyday sounds. This involves exposure to audio tapes and sounds related to their daily life, including voices of family and friends, snippets of favorite songs, and sounds associated with past work or leisure activities. The control group will undergo a program called Intensive Sensorial Emotional Stimulation (ISES), matching the frequency, intensity, and session duration of the experimental group but without Neurowave system utilization. Distinctively, the control group will not utilize Neurowave technology. Instead, they will follow a traditional rehabilitation approach incorporating paper materials, live photos, face-to-face interaction with the therapist, and the conventional listening of music tapes. This method aims to replicate an emotionally engaging environment, serving as a comparative reference to the experimental group's Neurowave-assisted experience.
  Interventions: Other: Intensive Sensorial Emotional Stimulation (ISES)

INTERVENTIONS:
Device: Intensive Neurowave Emotional Stimulation (INES) — Patients will undergo Neurowave-assisted multisensory stimulation five days a week for four weeks, featuring emotionally significant audio-visual content tied to personal history. Control group participants will experience primary auditory stimulation through familiar sounds, following a traditional rehabilitation approach mimicking the experimental group's frequency and intensity but without Neurowave use. This allows for a meaningful comparison of the two groups' experiences.
  Other Names: Intensive Sensorial Emotional Stimulation (ISES)
  Arms: Experimental group
Other: Intensive Sensorial Emotional Stimulation (ISES) — The Intensive Sensorial Emotional Stimulation (ISES) in the control group involves primary auditory stimulation with emotionally rich everyday sounds, including familiar voices, favorite songs, and sounds related to daily life and past activities. It mimics the experimental group's frequency and intensity, lasting 45 minutes per session, five days a week, for four weeks. Unlike the experimental group using Neurowave, the control group follows a traditional rehabilitation approach with paper materials, live photos, face-to-face interaction, and classic music tapes, facilitating a meaningful comparison between the two groups' experiences.
  Other Names: traditional rehabilitation
  Arms: Control group

SUMMARY:
This is a randomized and controlled pilot study investigating the effects of intensive emotional stimulation with neurological waves (INES) on cognitive-motor functions in patients diagnosed with Vegetative State (VS) and Minimally Conscious State (MCS) following severe brain injury. The study aims to enroll at least 20 patients aged between 18 and 65 over 18 months. Patients will be recruited from the Neurorehabilitation Unit of Piedmont Hospital, IRCCS Centro Neurolesi Bonino Pulejo in Messina. The experimental group will receive multisensory stimulation using Neurowave (INES) for four weeks, five days a week, 45 minutes per session. The control group will undergo a traditional multisensory stimulation program.

Enrollment will use simple random sampling to minimize bias. Caregivers will provide biographical information, and both groups will be monitored using event-related potentials. Clinical scales will evaluate cognitive-motor outcomes at different time points. The study includes a one-month follow-up to assess long-term results. Data will be collected and exported for statistical analysis.

DETAILED DESCRIPTION:
This study aims to investigate the cognitive-motor effects of emotionally significant advanced multisensory stimulation (INES) in patients diagnosed with Vegetative State (VS) and Minimally Conscious State (MCS) following severe acquired brain injury. Primary objectives include exploring short- and long-term efficacy through clinical-psychometric follow-up and examining potential correlations between neurophysiological and clinical-psychometric parameters as predictive indices of recovery.

The secondary objectives concern the implementation of highly specialized technological innovations in current clinical practice, and evaluating the rehabilitation effectiveness of advanced treatment with Neurological Waves.

Therefore, the study aims to develop models and protocols for multisensory rehabilitation stimulation and evaluate the synergies between different stimulation modalities and advanced cognitive electrophysiology techniques. Furthermore, the research aims to promote clinical investigations and systematic monitoring of post-acute patients, focusing on the quantitative analysis of EEG and Cognitive Evoked Potentials to unconventional sensory stimuli with emotionally significant content. The study also deepens the understanding of the role of the metabolic-nutritional state in the cognitive-motor recovery of patients with disorders of consciousness.

The present study is a randomized controlled pilot study, with an interventional, non-pharmacological, and single-center design.

Materials and methods:

The study will consecutively enroll at least 20 adult subjects diagnosed with disorders of consciousness at the Neurorehabilitation Unit of the Piedmont Hospital. Comprehensive multidimensional assessments will be conducted at baseline (T0), followed by an intensive one-month course of advanced multisensory training using Neurowave (INES) for the experimental group and conventional multisensory stimulation (ISES) for the control group. Evaluation at the end of each training cycle (T1) and a one-month follow-up (T2) will provide information on long-term results.

Inclusion criterion:

Participants must be between the ages of 18 and 65, with a Glasgow Coma Scale (GCS) score greater than 8 and a Cognitive Scale Level (LCF) between 1 and 3. Informed consent must be obtained from their legal guardian.

Exclusion criteria:

Exclusion criteria include individuals outside the specified age range, lack of legal guardian consent, anatomical alterations that prevent the correct placement of electrodes, and absence of neurophysiological responses in visual and auditory evoked potentials.

Registration start and end dates:

The study implementation period is expected to be from December 2023 to March 2025, with a total study duration of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Glasgow Coma Scale (GCS) > 8.
* Level of Cognitive Scale (LCF) = 1-3.
* Consent is signed by the legal guardian.

Exclusion Criteria:

* Age < 18 years or > 65 years.
* Lack of consent from the legal guardian.
* Patients with cranial anatomical alterations hindering proper electrode, headset, etc., placement.
* Patients showed no neurophysiological responses in visual evoked potentials (VEP) and no V wave in auditory evoked potentials (AEP).

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-12-14 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Cognitive-Motor Functional Improvement Score | clinical and psychometric scales will be administered to patients before starting sensory stimulation treatment (time T0), at the end of the stimulation cycle after 4 weeks (time T1), and one month after T1 (follow-up - Time T2).
  The "Cognitive-Motor Functional Improvement Score" is a composite index designed to assess the enhancement of cognitive and motor functions in study participants. This score takes into account various clinical and psychometric measurements, including parameters such as the Glasgow Coma Scale (GCS), the Glasgow Outcome Scale (GOS), the Level of Cognitive Functioning (LCF), the Coma Recovery Scale-Revised (CRS-R), the Disability Rating Scale (DRS), and the Functional Communication Scale (FCS). The score reflects the progression in cognitive and motor abilities of patients before, during, and after the treatment, providing a comprehensive measure of the success of the rehabilitation intervention.
Examine Short and Long-Term Efficacy | clinical and psychometric scales will be administered to patients before starting sensory stimulation treatment (time T0), at the end of the stimulation cycle after 4 weeks (time T1), and one month after T1 (follow-up - Time T2).
  Examine the correlation between neurophysiological and clinical-psychometric parameters to monitor the long-term cognitive-motor effects of advanced multisensory training in individuals with disorders of consciousness, identifying potential predictive indices of recovery. Assessment Method: Clinical evaluations and psychometric tests focusing on cognitive-motor, neurophysiological, and metabolic-nutritional outcomes. Timing: Short-term assessments post-training (T1) and long-term follow-up one month after treatment completion (T2).

SECONDARY OUTCOMES:
Study Neurophysiological and Clinical Correlations | clinical and psychometric scales will be administered to patients before starting sensory stimulation treatment (time T0), at the end of the stimulation cycle after 4 weeks (time T1), and one month after T1 (follow-up - Time T2).
  The comprehensive evaluation includes continuous clinical monitoring, electroencephalographic (EEG) assessments, and metabolic-nutritional evaluations. The goal is to establish meaningful correlations contributing to predictive indices for long-term cognitive-motor recovery in individuals with consciousness disorders. Evaluation: Clinical Monitoring: Continuous assessment of clinical and psychometric parameters. Electroencephalographic (EEG) Assessments: Recording and analysis of EEG data to monitor neurophysiological responses.
  Timing: Pre-treatment (T0): Baseline assessment before the commencement of advanced multisensory training. Post-treatment (T1): Evaluation immediately after the completion of the training program.
  Follow-up (T2): Long-term assessment one month after the conclusion of the treatment to gauge sustained effects and correlations.
Explore the Role of Metabolic-Nutritional Status | clinical and psychometric scales will be administered to patients before starting sensory stimulation treatment (time T0), at the end of the stimulation cycle after 4 weeks (time T1), and one month after T1 (follow-up - Time T2).
  This outcome measure investigates the influence of metabolic-nutritional status on cognitive-motor recovery in patients with consciousness disorders. Through a specialized early assessment, it aims to deepen our understanding of how factors such as BMI, creatinine/height, albumin, total proteins, and lymphocyte count contribute to the overall recovery process. The study seeks to unravel the intricate interplay between metabolic-nutritional health and cognitive-motor outcomes in individuals undergoing advanced multisensory training, providing valuable insights for tailored interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia Maggio, Principal Investigator — IRCCS Centro Neurolesi Bonino Pulejo
Locations (1):
- IRCCS Centro Neurolesi Bonino Pulejo, Messina, Italy/Messina, Italy

IPD SHARING:
Plan to Share IPD: No
We plan to make individual participant data (IPD) available to other researchers. This means that we intend to publish the databases, allowing access for other researchers to utilize the individualized data collected from each participant in our study. By doing so, we aim to contribute to the broader scientific community, fostering collaboration and enabling further exploration and analysis of the information gathered during our research.

REFERENCES:
- [Result] Sergent C, Faugeras F, Rohaut B, Perrin F, Valente M, Tallon-Baudry C, Cohen L, Naccache L. Multidimensional cognitive evaluation of patients with disorders of consciousness using EEG: A proof of concept study. Neuroimage Clin. 2016 Dec 10;13:455-469. doi: 10.1016/j.nicl.2016.12.004. eCollection 2017. PMID 28116238
- [Result] Padilla R, Domina A. Effectiveness of Sensory Stimulation to Improve Arousal and Alertness of People in a Coma or Persistent Vegetative State After Traumatic Brain Injury: A Systematic Review. Am J Occup Ther. 2016 May-Jun;70(3):7003180030p1-8. doi: 10.5014/ajot.2016.021022. PMID 27089287
- [Result] Lombardi F, Taricco M, De Tanti A, Telaro E, Liberati A. Sensory stimulation for brain injured individuals in coma or vegetative state. Cochrane Database Syst Rev. 2002;2002(2):CD001427. doi: 10.1002/14651858.CD001427. PMID 12076410
- [Result] Keller I, Hulsdunk A, Muller F. The influence of acoustic and tactile stimulation on vegetative parameters and EEG in persistent vegetative state. Funct Neurol. 2007 Jul-Sep;22(3):159-63. PMID 17925166